CLINICAL TRIAL: NCT04249622
Title: Phase II Trial of Rifaximin in Patients With Early Stage HER2 Positive Breast Cancer With Gastrointestinal Toxicities Related to Pertuzumab-Based Therapy
Brief Title: Rifaximin for the Treatment of Gastrointestinal Toxicities Related to Pertuzumab-Based Therapy in Patients With Stage I-III HER2 Positive Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow accrual
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MC18C3; NCI-2020-00332 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC18C3 (Other: Mayo Clinic in Florida); 18-009108 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2020-01-27; First posted 2020-01-31 (Actual); Results first posted 2025-08-07 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-08

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage IA Breast Cancer AJCC v8; Anatomic Stage IB Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage IIA Breast Cancer AJCC v8; Anatomic Stage IIB Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Anatomic Stage IIIB Breast Cancer AJCC v8; Anatomic Stage IIIC Breast Cancer AJCC v8; HER2 Positive Breast Carcinoma; Prognostic Stage I Breast Cancer AJCC v8; Prognostic Stage IA Breast Cancer AJCC v8; Prognostic Stage IB Breast Cancer AJCC v8; Prognostic Stage II Breast Cancer AJCC v8; Prognostic Stage IIA Breast Cancer AJCC v8; Prognostic Stage IIB Breast Cancer AJCC v8; Prognostic Stage III Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8; Prognostic Stage IIIB Breast Cancer AJCC v8; Prognostic Stage IIIC Breast Cancer AJCC v8
MeSH Terms: interventions — Practice Guidelines as Topic; Standard of Care; Rifaximin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (rifaximin, pertuzumab-based chemotherapy) (Experimental): Patients that experience PIGT after receiving first standard of care cycle of pertuzumab-based chemotherapy receive rifaximin PO BID on days 1-5 and standard of care pertuzumab-based chemotherapy on day 1. Treatment repeats every 21 days for up to 5 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Best Practice; Other: Questionnaire Administration; Drug: Rifaximin
- Arm II (pertuzumab-based chemotherapy) (Active Comparator): Patients that do not experience PIGT after receiving first standard of care cycle of pertuzumab-based chemotherapy continue receiving standard of care pertuzumab-based chemotherapy on day 1. Treatment repeats every 21 days for up to 5 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Best Practice; Other: Questionnaire Administration

INTERVENTIONS:
Other: Best Practice — Given standard of care pertuzumab-based chemotherapy
  Other Names: standard of care; standard therapy
Other: Questionnaire Administration — Ancillary studies
Drug: Rifaximin — Given PO
  Other Names: Xifaxan
  Arms: Arm I (rifaximin, pertuzumab-based chemotherapy)

SUMMARY:
This phase II trial studies how well rifaximin works for the treatment of gastrointestinal toxicities related to pertuzumab-based therapy in patients with stage I-III HER2 positive breast cancer. Rifaximin may reduce the incidence and severity of pertuzumab induced gastrointestinal toxicities without interrupting or delaying the chemotherapy schedule.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the reduction rate of grade >= 2 abdominal toxicities, including abdominal distension, abdominal pain, diarrhea, dyspepsia, stomach pain, and typhlitis according to the National Cancer Institute Common Terminology for Adverse Events version 5.0 (NCI CTCAE v5.0) with the use of rifaximin in stage II-III HER-2 positive breast cancer patients with pertuzumab induced gastrointestinal toxicities.

SECONDARY OBJECTIVES:

I. Evaluate dose reductions, dose delays and discontinuation of treatment with pertuzumab due to gastrointestinal side effects.

II. Evaluate and measure the change in the Bristol stool scale before and after rifaximin treatment.

III. Evaluate and measure the change in the 4-point Likert scale patient questionnaire before and after rifaximin treatment.

CORRELATIVE STUDY OBJECTIVES:

I. Evaluate changes in the fecal microbiome, hydrogen breath test, and permeability test before and after rifaximin.

II. Evaluate changes in the fecal microbiome, hydrogen breath test, and permeability test before and after pertuzumab-based chemotherapy.

III. Evaluate the difference in the fecal microbiome, hydrogen breath test, and permeability test among patients with or without pertuzumab induced gastrointestinal toxicities (PIGT).

OUTLINE: Patients are assigned to 1 of 2 arms.

ARM I (GRADE >= 2 PIGT): Patients that experience PIGT after receiving first standard of care cycle of pertuzumab-based chemotherapy receive rifaximin orally (PO) twice daily (BID) on days 1-5 and standard of care pertuzumab-based chemotherapy on day 1. Treatment repeats every 21 days for up to 5 cycles in the absence of disease progression or unacceptable toxicity.

ARM II (GRADE =< 1 PIGT): Patients that do not experience PIGT after receiving first standard of care cycle of pertuzumab-based chemotherapy continue receiving standard of care pertuzumab-based chemotherapy on day 1. Treatment repeats every 21 days for up to 5 cycles in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* PRE-REGISTRATION INCLUSION CRITERIA
* Age >= 18 years
* Histological confirmation of HER2 positive breast cancer stage I-III per American Joint Committee on Cancer (AJCC) staging 8th edition
* Provide written informed consent
* Breast cancer patients who will be receiving pertuzumab-based chemotherapy with either TCHP (docetaxel, carboplatin, trastuzumab, and pertuzumab) or docetaxel/paclitaxel, trastuzumab, and pertuzumab
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1, or 2
* Hemoglobin >= 10.0 g/dL (obtained =< 30 days prior to pre-registration)
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L (obtained =< 30 days prior to pre-registration)
* Platelet count >= 100 x 10^9/L (obtained =< 30 days prior to pre-registration)
* Total bilirubin =< 1.5 x ULN (institutional upper limit of normal) (obtained =< 30 days prior to pre-registration)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x ULN (obtained =< 30 days prior to pre-registration)
* Serum or plasma creatinine =< 1.5 x ULN (obtained =< 30 days prior to pre-registration)
* Calculated creatinine clearance >= 45 ml/min using the Cockcroft-Gault formula (obtained =< 30 days prior to pre-registration)
* Negative serum pregnancy test done =< 30 days prior to pre-registration, for person of childbearing potential only
* Willingness to return to enrolling institution for follow-up (during the active monitoring phase of the study)
* Willingness to provide mandatory stool specimen for correlative research
* Ability to complete questionnaire(s) by themselves or with assistance
* REGISTRATION INCLUSION CRITERIA
* Received pertuzumab based regimens in the adjuvant or neoadjuvant setting
* Hemoglobin >= 8.0 g/dL (obtained =< 14 days prior to registration)
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L (obtained =< 14 days prior to registration)
* Platelet count >= 100 x 10^9/L (obtained =< 14 days prior to registration)
* Total bilirubin =< 1.5 x ULN (institutional upper limit of normal) (obtained =< 14 days prior to registration)
* AST (SGOT)/ALT (SGPT) =< 2.5 x ULN (obtained =< 14 days prior to registration)
* Serum or plasma creatinine =< 1.5 x ULN (obtained =< 14 days prior to registration)
* Calculated creatinine clearance >= 45 ml/min using the Cockcroft-Gault formula (obtained =< 14 days prior to registration)

Exclusion Criteria:

* PRE-REGISTRATION EXCLUSION CRITERIA
* History of myocardial infarction =< 6 months prior to pre-registration, or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias
* Failure to recover from acute, reversible effects of prior therapy regardless of interval since last treatment

  * EXCEPTION: Grade 1 peripheral (sensory) neuropathy that has been stable for at least 3 months since completion of prior treatment
* Uncontrolled intercurrent non-cardiac illness including, but not limited to:

  * Ongoing or active infection
  * Psychiatric illness/social situations
  * Dyspnea at rest due to complications of advanced malignancy or other disease that requires continuous oxygen therapy
  * Any other conditions that would limit compliance with study requirements
* Immunocompromised patients and patients known to be human immunodeficiency virus (HIV) positive and currently receiving antiretroviral therapy

  * NOTE: Patients known to be HIV positive, but without clinical evidence of an immunocompromised state, are eligible for this trial
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm (adjust to protocol if applicable)
* Any of the following because this study involves an agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown

  * Pregnant women
  * Nursing women
  * Women of childbearing potential who are unwilling to employ adequate contraception
* Current colostomy or ileostomy
* History of inflammatory bowel disease
* History of irritable bowel syndrome
* History of arteriovenous malformations
* History of gastrointestinal bleeds
* Previous surgical resection of the small bowel or colon
* Previous allergy to rifaximin or its derivatives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-09-18 (Actual); Primary Completion 2022-12-27 (Actual); Study Completion 2022-12-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saranya Chumsri, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (Rifaximin, Pertuzumab-based Chemotherapy): Patients that experience PIGT after receiving first standard of care cycle of pertuzumab-based chemotherapy receive rifaximin PO BID on days 1-5 and standard of care pertuzumab-based chemotherapy on day 1. Treatment repeats every 21 days for up to 5 cycles in the absence of disease progression or unacceptable toxicity.>
  * Best Practice: Given standard of care pertuzumab-based chemotherapy >
  * Questionnaire Administration: Ancillary studies >
  * Rifaximin: Given PO
- Arm II (Pertuzumab-based Chemotherapy): Patients that do not experience PIGT after receiving first standard of care cycle of pertuzumab-based chemotherapy continue receiving standard of care pertuzumab-based chemotherapy on day 1. Treatment repeats every 21 days for up to 5 cycles in the absence of disease progression or unacceptable toxicity.>
  * Best Practice: Given standard of care pertuzumab-based chemotherapy >
  * Questionnaire Administration: Ancillary studies
Period: Overall Study
Arm/Group | Arm I (Rifaximin, Pertuzumab-based Chemotherapy) | Arm II (Pertuzumab-based Chemotherapy)
Started | 18 | 2
Completed | 15 | 1
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Alternative therapy | 1 | 0
Not completed — Discontinuation of pertuzumab | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm II (Pertuzumab-based Chemotherapy): Patients that do not experience PIGT after receiving first standard of care cycle of pertuzumab-based chemotherapy continue receiving standard of care pertuzumab-based chemotherapy on day 1. Treatment repeats every 21 days for up to 5 cycles in the absence of disease progression or unacceptable toxicity.>
  * Best Practice: Given standard of care pertuzumab-based chemotherapy>
  * Questionnaire Administration: Ancillary studies
- Total: Total of all reporting groups
Arm/Group | Arm I (Rifaximin, Pertuzumab-based Chemotherapy) | Arm II (Pertuzumab-based Chemotherapy) | Total
Number analyzed (Participants) | 18 | 2 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.8 (9.72) | 55.0 (7.07) | 53.9 (9.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 2 | 20
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 16 | 2 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 18 | 2 | 20
ECOG Performance Status [Count of Participants; unit: Participants] — 0 Fully active, able to carry on all pre-disease performance without restriction>
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work>
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours>
  3. Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours>
  4. Completely disabled; cannot carry on any selfcare; totally confined to bed or chair>
  5. Dead
  Participants
    0 | 16 | 2 | 18
    1 | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Reduction Rate of >= Grade 2 Abdominal Toxicities Including Abdominal Distension, Abdominal Pain, Diarrhea, Dyspepsia, Stomach Pain, and Typhlitis
Description: Based on the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. The proportion of successes will be estimated by the number of successes divided by the total number of evaluable patients. Confidence intervals for the true success proportion will be calculated according to the approach of Duffy and Santner (1987).
Time Frame: Through study completion (approximately 2 years, 3 months)
Population: Only patients that received rifaximin were included in analysis
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm I (Rifaximin, Pertuzumab-based Chemotherapy)
Number analyzed (Participants) | 18
proportion of participants | 0.833 [0.5858 to 0.9642]

2. Secondary Outcome: Dose Reductions of Treatment With Pertuzumab
Description: Number of patients that experienced a dose reductions with pertuzumab due to gastrointestinal side effects.
Time Frame: Up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Rifaximin, Pertuzumab-based Chemotherapy) | Arm II (Pertuzumab-based Chemotherapy)
Number analyzed (Participants) | 18 | 2
Participants | 10 | 0

3. Secondary Outcome: Dose Delays of Treatment With Pertuzumab
Description: Number of patients that experienced a dose delay with pertuzumab due to gastrointestinal side effects.
Time Frame: Up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Rifaximin, Pertuzumab-based Chemotherapy) | Arm II (Pertuzumab-based Chemotherapy)
Number analyzed (Participants) | 18 | 2
Participants | 1 | 0

4. Secondary Outcome: Discontinuation of Treatment With Pertuzumab
Description: The number of patients that experienced discontinuation of treatment with pertuzumab due to gastrointestinal side effects.
Time Frame: Up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Rifaximin, Pertuzumab-based Chemotherapy) | Arm II (Pertuzumab-based Chemotherapy)
Number analyzed (Participants) | 18 | 2
Participants | 0 | 0

5. Secondary Outcome: Number of Patient With a Reduction of Mean Number of Stools
Description: Number of patients that experienced a reduction of mean number of stools recorded while on treatment compared to baseline will be reported
Time Frame: Up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Rifaximin, Pertuzumab-based Chemotherapy) | Arm II (Pertuzumab-based Chemotherapy)
Number analyzed (Participants) | 18 | 2
Participants | 7 | 0

6. Secondary Outcome: Average Maximum Pertuzumab Induced Gastrointestinal Toxicities (PIGT) Score
Description: Maximum PIGT score represents the maximum grade of adverse event experienced by a patient out of all gastrointestinal adverse events. PIGT scores are assessed according to NCI CTCAE v5.0, with a minimum grade of 0 (no event) and maximum grade of 5 (death).
Time Frame: Baseline (at enrollment); following each treatment cycle (21 days +/- 7 days), up to 5 cycles
Population: Only patients in arm 1 were included in analysis. Patients in arm 2 did not experience PIGT. Only patients still on treatment were included in each cycle's analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm I (Rifaximin, Pertuzumab-based Chemotherapy) | Arm II (Pertuzumab-based Chemotherapy)
Number analyzed (Participants) | 18 | 0
units on a scale
  Baseline | 2.17 (0.38) |
  Cycle 1 | 1.61 (0.78) |
  Cycle 2 | 1.83 (0.79) |
  Cycle 3: number analyzed (Participants) | 17 | 0
  Cycle 3 | 1.71 (0.85) |
  Cycle 4: number analyzed (Participants) | 16 | 0
  Cycle 4 | 1.5 (0.73) |
  Cycle 5: number analyzed (Participants) | 15 | 0
  Cycle 5 | 1.53 (0.74) |

7. Other Pre Specified Outcome: Changes in the Fecal Microbiome, Hydrogen Breath Test, and Permeability Test - Rifaximin
Description: Descriptive statistics (mean, standard deviation [sd], median, interquartile range [iqr]) and longitudinal plots (raw value, change, change in percentage) will be used to summarize the baseline levels of hydrogen/methane peak by hydrogen breath test , diversity of gut microbiome(number of species) and specific species by fecal microbiome, and levels of urine mannitol and lactulose by permeability test before and after rifaximin.
Time Frame: Baseline up to 3 years
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Changes in the Fecal Microbiome, Hydrogen Breath Test, and Permeability Test - Pertuzumab
Description: Descriptive statistics (mean, sd, median, iqr) and longitudinal plots (raw value, change, change in percentage) will be used to summarize the baseline levels of hydrogen/methane peak by hydrogen breath test, diversity of gut microbiome (number of species) and specific species by fecal microbiome, and levels of urine mannitol and lactulose by permeability test before and after pertuzumab-based chemotherapy.
Time Frame: Baseline up to 3 years
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Difference in the Fecal Microbiome, Hydrogen Breath Test, and Permeability Test
Description: Descriptive statistics (mean, sd, median, iqr) and longitudinal plots (raw value, change, change in percentage) will be used to the fecal microbiome, hydrogen breath test, and permeability test among patients with or without PIGT. The study is not powered to detect any differences between the two arms; the main purpose is to quantify and evaluate differences descriptively between patients who develop and do not develop PIGT (between arm 1 and arm 2) to inform subsequent research.
Time Frame: Up to 3 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 3 years
Groups:
- Arm I (Rifaximin, Pertuzumab-based Chemotherapy): Patients that experience PIGT after receiving first standard of care cycle of pertuzumab-based chemotherapy receive rifaximin PO BID on days 1-5 and standard of care pertuzumab-based chemotherapy on day 1. Treatment repeats every 21 days for up to 5 cycles in the absence of disease progression or unacceptable toxicity. >
  * Best Practice: Given standard of care pertuzumab-based chemotherapy >
  * Questionnaire Administration: Ancillary studies >
  * Rifaximin: Given PO
- Arm II (Pertuzumab-based Chemotherapy): Patients that do not experience PIGT after receiving first standard of care cycle of pertuzumab-based chemotherapy continue receiving standard of care pertuzumab-based chemotherapy on day 1. Treatment repeats every 21 days for up to 5 cycles in the absence of disease progression or unacceptable toxicity. > > Best Practice: Given standard of care pertuzumab-based chemotherapy >
  > Questionnaire Administration: Ancillary studies
Arm/Group | Arm I (Rifaximin, Pertuzumab-based Chemotherapy) | Arm II (Pertuzumab-based Chemotherapy)
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/2
Serious Adverse Events (participants affected / at risk) | 1/18 | 0/2
Other Adverse Events (participants affected / at risk) | 18/18 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Rifaximin, Pertuzumab-based Chemotherapy) (N=18) | Arm II (Pertuzumab-based Chemotherapy) (N=2)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Rifaximin, Pertuzumab-based Chemotherapy) (N=18) | Arm II (Pertuzumab-based Chemotherapy) (N=2)
Anemia (Blood and lymphatic system disorders) | 16 (67) | 2 (6)
Blood and lymph sys disorders - Oth Spec (Blood and lymphatic system disorders) | 4 (6) | 0 (0)
Cardiac disorders - Other, specify (Cardiac disorders) | 2 (3) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 4 (15) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Blurred vision (Eye disorders) | 5 (14) | 0 (0)
Dry eye (Eye disorders) | 6 (15) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 2 (3) | 0 (0)
Watering eyes (Eye disorders) | 0 (0) | 1 (4)
Constipation (Gastrointestinal disorders) | 6 (20) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 17 (67) | 2 (6)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4 (11) | 1 (5)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 7 (12) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 2 (9) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 14 (43) | 2 (6)
Rectal hemorrhage (Gastrointestinal disorders) | 2 (7) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (5) | 0 (0)
Chills (General disorders) | 1 (2) | 0 (0)
Edema limbs (General disorders) | 3 (3) | 0 (0)
Fatigue (General disorders) | 14 (55) | 2 (6)
Fever (General disorders) | 1 (1) | 0 (0)
Gen disord and admin site conds-Oth spec (General disorders) | 7 (23) | 1 (3)
Pain (General disorders) | 0 (0) | 1 (1)
Infections and infestations - Oth spec (Infections and infestations) | 3 (4) | 0 (0)
Papulopustular rash (Infections and infestations) | 1 (4) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Thrush (Infections and infestations) | 1 (3) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 8 (25) | 2 (5)
Alkaline phosphatase increased (Investigations) | 3 (4) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 4 (8) | 1 (2)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 2 (5) | 1 (4)
Creatinine increased (Investigations) | 1 (1) | 0 (0)
Investigations - Other, specify (Investigations) | 4 (11) | 2 (2)
Lymphocyte count decreased (Investigations) | 4 (7) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (7) | 0 (0)
Platelet count decreased (Investigations) | 8 (18) | 0 (0)
White blood cell decreased (Investigations) | 2 (6) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (5) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperphosphatemia (Metabolism and nutrition disorders) | 2 (4) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (7) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 11 (25) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 8 (22) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Metabolism, nutrition disord - Oth spec (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (6) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 7 (17) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal, conn tissue - Oth spec (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (10) | 1 (2)
Dizziness (Nervous system disorders) | 13 (32) | 1 (4)
Dysgeusia (Nervous system disorders) | 8 (32) | 0 (0)
Headache (Nervous system disorders) | 9 (23) | 2 (4)
Nervous system disorders - Oth spec (Nervous system disorders) | 5 (11) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (3) | 1 (4)
Peripheral sensory neuropathy (Nervous system disorders) | 4 (15) | 1 (5)
Presyncope (Nervous system disorders) | 1 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (10) | 0 (0)
Renal and urinary disorders - Oth spec (Renal and urinary disorders) | 1 (1) | 0 (0)
Dyspareunia (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (5) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (7) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (5) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 4 (9) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 2 (5) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 12 (47) | 1 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (13) | 1 (3)
Rash acneiform (Skin and subcutaneous tissue disorders) | 3 (10) | 1 (5)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 (16) | 0 (0)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 4 (6) | 0 (0)
Telangiectasia (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
Hot flashes (Vascular disorders) | 1 (3) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-27): https://cdn.clinicaltrials.gov/large-docs/22/NCT04249622/Prot_SAP_000.pdf
  • Informed Consent Form (2021-12-29): https://cdn.clinicaltrials.gov/large-docs/22/NCT04249622/ICF_001.pdf